CLINICAL TRIAL: NCT02917811
Title: Red Cell Distribution Width (RDW) as a Prognostic Marker in ICU
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, MD, Università degli Studi di Ferrara
Other Study IDs: 20042016
Record Dates: First submitted 2016-09-13; First posted 2016-09-28 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Blood Transfusion; Biochemical Marker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ICU patients

SUMMARY:
The aim of this study is to verify if high values of RDW are useful prognostic marker for ICU mortality and 90-days mortality. Moreover, we will investigate the prognostic value of RDW in specific subgroup population with some clinical characteristic wich may modify RDW baseline values, i.e. transfused patients or patients with high markers of hemolysis

ELIGIBILITY:
Inclusion Criteria:

* Unselected ICU patients

Exclusion Criteria:

* Length of stay in ICU <48 hours
* Hematological disease
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to ICU will be considered for the study
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
90-days mortality | 90 days

SECONDARY OUTCOMES:
ICU mortality | 90 days
Length of mechanical ventilation | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sant'Anna Hospital, Ferrara, Ferrara, Italy

REFERENCES:
- [Result] Kim CH, Park JT, Kim EJ, Han JH, Han JS, Choi JY, Han SH, Yoo TH, Kim YS, Kang SW, Oh HJ. An increase in red blood cell distribution width from baseline predicts mortality in patients with severe sepsis or septic shock. Crit Care. 2013 Dec 9;17(6):R282. doi: 10.1186/cc13145. PMID 24321201
- [Result] Lorente L, Martin MM, Abreu-Gonzalez P, Sole-Violan J, Ferreres J, Labarta L, Diaz C, Gonzalez O, Garcia D, Jimenez A, Borreguero-Leon JM. Red blood cell distribution width during the first week is associated with severity and mortality in septic patients. PLoS One. 2014 Aug 25;9(8):e105436. doi: 10.1371/journal.pone.0105436. eCollection 2014. PMID 25153089